CLINICAL TRIAL: NCT04278456
Title: The Effect of the Anesthesia Modality Used in Women Giving Birth Under Caesarian Section on Postpartum Depression and/or Postoperative Melatonin Levels
Brief Title: Postpartum Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, REMZIYE AYSENUR NALBANT, MD, Erzincan University
Other Study IDs: EBYU 88
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Postpartum Depression; Melatonin
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- general anesthesia: c-section with general anesthesia
  Interventions: Behavioral: postpartum depression
- spinal anesthesia: c-section with spinal anesthesia
  Interventions: Behavioral: postpartum depression
- epidural anesthesia: c-section with epidural anesthesia
  Interventions: Behavioral: postpartum depression

INTERVENTIONS:
Behavioral: postpartum depression — melatonin levels in c-sections with different anesthesia modalities.

SUMMARY:
Our aim was to diagnose and initiate early treatment for postpartum depression by detecting the changes of melatonin levels in c-sections with different antesthesia modalities.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women c-section (using general or regional anesthesia) aged between 18-45 years

Exclusion Criteria:

* age under 18 or above 45, history of smoking, a diagnosis with mental retardation, psychiatric patients, use of antipsychotics or antidepressants, patients with sleeping disorders, hormone replacement theraphy patients.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — aged between 18-45 years
Study Population: pregnant women that will give birth by c-section (using general or regional anesthesia) aged between 18-45 years will be included to our study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-21 (Estimated); Primary Completion 2020-05-21 (Estimated); Study Completion 2020-07-21 (Estimated)

PRIMARY OUTCOMES:
edinburgh depression scale | 5 months
  below 12 is associated with depression

CONTACTS AND LOCATIONS:
Overall Officials: Remziye Ayşenur NALBANT, Principal Investigator — ERZİNCAN
Locations (1):
- Erzincan Byu, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andersen LP, Werner MU, Rosenberg J, Gogenur I. A systematic review of peri-operative melatonin. Anaesthesia. 2014 Oct;69(10):1163-71. doi: 10.1111/anae.12717. Epub 2014 May 19. PMID 24835540
- [Result] Maitra S, Baidya DK, Khanna P. Melatonin in perioperative medicine: Current perspective. Saudi J Anaesth. 2013 Jul;7(3):315-21. doi: 10.4103/1658-354X.115316. PMID 24015137
- [Result] Dianatkhah M, Ghaeli P, Hajhossein Talasaz A, Karimi A, Salehiomran A, Bina P, Jalali A, Ghaffary S, Shahmansouri N, Vejdani S. Evaluating the Potential Effect of Melatonin on the post-Cardiac Surgery Sleep Disorder. J Tehran Heart Cent. 2015 Jul 3;10(3):122-8. PMID 26697084